CLINICAL TRIAL: NCT03820492
Title: Multimodality Assessment of Intermediate Left Main Stenosis: Comparison of Optical Coherence Tomography-derived Minimal Lumen Area, Invasive Fractional Flow Reserve and FFRCT
Brief Title: Comparison of Optical Coherence Tomography-derived Minimal Lumen Area, Invasive Fractional Flow Reserve and FFRCT
Acronym: OPTICO-LM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OPTICO-LM
Record Dates: First submitted 2019-01-17; First posted 2019-01-29 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Coronary Stenosis
Keywords: Coronary artery disease; Fractional flow reserve; Optical coherence tomography; Computed tomography angiography
MeSH Terms: conditions — Coronary Stenosis; Coronary Artery Disease | interventions — Tomography, Optical Coherence; Computed Tomography Angiography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient with left-main stenosis (Other): Multimodality assessment of intermediate left main stenosis: Comparison of optical coherence tomography-derived minimal lumen area, invasive fractional flow reserve and FFRCT
  Interventions: Diagnostic Test: OCT, FFR, CTA and FFRCT

INTERVENTIONS:
Diagnostic Test: OCT, FFR, CTA and FFRCT — Multimodality assessment of intermediate left main stenosis: Comparison of optical coherence tomography-derived minimal lumen area, invasive fractional flow reserve and FFRCT

SUMMARY:
Significant left main (LM) stenosis is associated with a poor prognosis, therefore, adequate judgement of the prognostic significance of LM stenosis is essential to improve patients' prognosis. Recently, fractional flow reserve (FFR) has become widespread practice and carries a Class Ia recommendation to assess functional significance of intermediate coronary stenosis in patients with stable angina. Intravascular ultrasound (IVUS)-derived minimum lumen area (MLA) represents an accurate measure to determine LM significance as shown in multiple studies, while optical coherence tomography (OCT) ,which is a novel intracoronary imaging method with a greater spatial resolution (15μm vs. 100μm), faster image acquisition and facilitated image interpretation, OCT derived-MLA has never been validated against FFR and accordingly, it is not mentioned in the current guidelines for myocardial revascularization. Coronary computed tomography angiography (CTA) has emerged as a noninvasive alternative of coronary angiography with its excellent negative predictive value, while the positive predictive value of CTA is limited. Computational fluid dynamics is an emerging method that enables prediction of blood flow in coronary arteries and calculation of FFR from computed tomography (FFRCT) noninvasively. Noninvasive and accurate assessment of functional significance would bring a great benefit for patients with LM stenosis, however, there are no data to evaluate the diagnostic accuracy of FFRCT for LM stenosis in comparison with FFR and minimal lumen area derived by OCT.

This study will investigate the optimal OCT-derived MLA cut-off point and the diagnostic performance of FFRCT for intermediate LM stenosis compared with FFR ≤0.8 as a reference standard.

ELIGIBILITY:
Inclusion Criteria:

* Unprotected LM lesion [midshaft, and distal bifurcation (Medina 1,1,1 or 1,1,0 or 1,0,1 or 1,0,0)] of 30% to 80% angiographic diameter stenosis (DS) on visual estimation or equivocal disease by angiography.
* Age ≥18 years.
* Ability to give preliminary oral consent witnessed by an independent physician or sign written informed consent prior to any study-specific procedures.

Exclusion Criteria:

* Significant distal lesions (>50% angiographic DS on visual estimation within the left anterior descending artery [LAD] or left circumflex artery [LCX], except for ostium of LAD or LCX or diseased side branch [e.g. diagonal branch, obtuse marginal branch])
* Ostial LM disease.
* Acute coronary syndrome (ACS) (non-ST-elevation ACS and ST-elevation MI).
* LM In-stent restenosis.
* Previous coronary stenting of the left coronary system.
* Chronic total occlusion.
* Previous coronary artery bypass graft.
* Previous MI related to the left coronary artery.
* Occurrence of ventricularization or hypotension during engagement of the LM ostial lesion.
* The presence of hemodynamic instability.
* Known renal insufficiency (serum creatinine >1.5mg/dL or receiving dialysis).
* Female of childbearing potential (age <50 years and last menstruation within the last 12 months), who did not undergo tubal ligation, ovariectomy or hysterectomy.
* Life expectancy less than 1 year.
* Contraindication or known allergy against protocol-required medications including heparin, iodinated contrast, β-blocker, nitroglycerin, and adenosine.
* Body mass index >35kg/m2.
* Complex congenital heart disease other than anomalous coronary origins alone.
* Ventricular septal defect.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2019-05-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
OCT vs. FFR | Measurement at Procedure/ Baseline Visit
  - The area under the curve of OCT-derived MLA for FFR≤0.8
OCT vs. FFR | Measurement at Procedure/ Baseline Visit
  -The optimal cut-off point of OCT-derived MLA from receiver-operator characteristics curves for FFR≤0.8
FFRCT vs. FFR | Measurement at Procedure/ Baseline Visit
  Diagnostic accuracy, sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of FFRCT≤0.8 for FFR≤0.8

SECONDARY OUTCOMES:
OCT vs. FFR, RFR, resting Pd/Pa, FFRCT, QFR | Measurement at Procedure/ Baseline Visit
  - The area under the curve and the optimal cut-off point of OCT-derived MLA from receiver-operator characteristics curves for FFR≤0.75, RFR≤0.89, resting Pd/Pa≤0.91, and FFRCT≤0.80 and QFR≤0.80
OCT vs. FFR, RFR, resting Pd/Pa, FFRCT | Measurement at Procedure/ Baseline Visit
  - Predictability of MLA, minimal lumen diameter, area stenosis, lesion length, eccentricity index, and plaque characteristics (plaque rupture, fibroatheroma, and calcification) for FFR ≤0.8, FFR≤0.75, RFR≤0.89, resting Pd/Pa≤0.91, and FFRCT≤0.80 and QFR≤0.80
OCT vs. FFR, RFR, resting Pd/Pa, FFRCT | Measurement at Procedure/ Baseline Visit
  - Correlation among OCT-derived MLA, FFR, RFR, resting Pd/Pa, and FFRCT and QFR
OCT vs. CTA | Measurement at Procedure/ Baseline Visit
  - Correlation between luminal diameter stenosis of CTA and OCT-derived MLA
OCT vs. CTA | Measurement at Procedure/ Baseline Visit
  - Diagnostic accuracy of plaque characteristics with presumed high risk characteristics including napkin ring sign, low attenuation plaque (<30HU), positive remodelling (remodelling index >1.1), and spotty calcium (<3mm) for thin and thick cap fibroatheroma by OCT.
Clinical endpoint at 1 year | 12 Month
  Death
Clinical endpoint at 1 year | 12 Month
  Myocardial infarction
Clinical endpoint at 1 year | 12 Month
  Target vessel myocardial infarction
Clinical endpoint at 1 year | 12 Month
  Target lesion revascularization
Clinical endpoint at 1 year | 12 Month
  Target vessel revascularization
Clinical endpoint at 1 year | 12 Month
  Any revascularization
Clinical endpoint at 1 year | 12 Month
  Stent thrombosis
Clinical endpoint at 1 year | 12 Month
  Stroke and transient ischemic attack
Clinical endpoint at 1 year | 12 Month
  Acute renal failure

CONTACTS AND LOCATIONS:
Overall Officials: Lorenz Raeber, Prof. MD PhD, Principal Investigator — Inselspital
Locations (13):
- France (3):
  - Centre Hospitalier Universitaire de Clermont-Ferrand, Clermont-Ferrand
  - Institute Mutualiste Montsouris, Paris
  - Centre Cardiologique du Nord, Saint-Denis
- Germany (2):
  - Universitätsklinikum Giessen Justus-Liebig Universität, Giessen, Hesse
  - Friedrich Alexander Universität (FAU) , Medizinische Klinik 2 , Kardiologie und Angiologie, Erlangen
- Japan (6):
  - Ageo Central General Hospital, Ageo
  - Gifu heart center, Gifu
  - Department of Cardiovascular Medicine Shinshu University School of Medicine, Nagano
  - Kansai Medical University,, Osaka
  - Medical Corporation Ouyuukai Tokorozawa Heart Center, Saitama
  - Sapporo Higashi Tokushukai Hospital, Sapporo
- Switzerland (2):
  - Inselspital, Bern
  - CHUV, Lausanne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Makikallio T, Holm NR, Lindsay M, Spence MS, Erglis A, Menown IB, Trovik T, Eskola M, Romppanen H, Kellerth T, Ravkilde J, Jensen LO, Kalinauskas G, Linder RB, Pentikainen M, Hervold A, Banning A, Zaman A, Cotton J, Eriksen E, Margus S, Sorensen HT, Nielsen PH, Niemela M, Kervinen K, Lassen JF, Maeng M, Oldroyd K, Berg G, Walsh SJ, Hanratty CG, Kumsars I, Stradins P, Steigen TK, Frobert O, Graham AN, Endresen PC, Corbascio M, Kajander O, Trivedi U, Hartikainen J, Anttila V, Hildick-Smith D, Thuesen L, Christiansen EH; NOBLE study investigators. Percutaneous coronary angioplasty versus coronary artery bypass grafting in treatment of unprotected left main stenosis (NOBLE): a prospective, randomised, open-label, non-inferiority trial. Lancet. 2016 Dec 3;388(10061):2743-2752. doi: 10.1016/S0140-6736(16)32052-9. Epub 2016 Oct 31. PMID 27810312
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Jasti V, Ivan E, Yalamanchili V, Wongpraparut N, Leesar MA. Correlations between fractional flow reserve and intravascular ultrasound in patients with an ambiguous left main coronary artery stenosis. Circulation. 2004 Nov 2;110(18):2831-6. doi: 10.1161/01.CIR.0000146338.62813.E7. Epub 2004 Oct 18. PMID 15492302
- [Background] de la Torre Hernandez JM, Hernandez Hernandez F, Alfonso F, Rumoroso JR, Lopez-Palop R, Sadaba M, Carrillo P, Rondan J, Lozano I, Ruiz Nodar JM, Baz JA, Fernandez Nofrerias E, Pajin F, Garcia Camarero T, Gutierrez H; LITRO Study Group (Spanish Working Group on Interventional Cardiology). Prospective application of pre-defined intravascular ultrasound criteria for assessment of intermediate left main coronary artery lesions results from the multicenter LITRO study. J Am Coll Cardiol. 2011 Jul 19;58(4):351-8. doi: 10.1016/j.jacc.2011.02.064. PMID 21757111
- [Background] Norgaard BL, Leipsic J, Gaur S, Seneviratne S, Ko BS, Ito H, Jensen JM, Mauri L, De Bruyne B, Bezerra H, Osawa K, Marwan M, Naber C, Erglis A, Park SJ, Christiansen EH, Kaltoft A, Lassen JF, Botker HE, Achenbach S; NXT Trial Study Group. Diagnostic performance of noninvasive fractional flow reserve derived from coronary computed tomography angiography in suspected coronary artery disease: the NXT trial (Analysis of Coronary Blood Flow Using CT Angiography: Next Steps). J Am Coll Cardiol. 2014 Apr 1;63(12):1145-1155. doi: 10.1016/j.jacc.2013.11.043. Epub 2014 Jan 30. PMID 24486266